CLINICAL TRIAL: NCT00944164
Title: Test the Feasibility of Primary Care Obesity Prevention and Treatment - Pilot Study
Brief Title: Primary Care Obesity Prevention and Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Group Health (Unknown); Fred Hutchinson Cancer Center (Other)
Responsible Party: Rona Levy, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-06-C40
Record Dates: First submitted 2009-07-09; First posted 2009-07-23 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Healthy; Exercise; Safety

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy eating/physical activity (Experimental)
  Interventions: Behavioral: Healthy eating and physical activity
- Safety/Injury prevention (Active Comparator)
  Interventions: Behavioral: Safety and injury prevention

INTERVENTIONS:
Behavioral: Healthy eating and physical activity — Parent counseling and coaching regarding healthy eating and physical activity habits for their child
  Arms: Healthy eating/physical activity
Behavioral: Safety and injury prevention — Parent counseling and coaching regarding general personal and household safety
  Arms: Safety/Injury prevention

SUMMARY:
The overall objective of this pilot is to demonstrate the feasibility of a low-cost intervention targeting obesity prevention among children in a primary care setting.

Specifically, the investigators aim to answer the following questions:

Can the investigators recruit and retain patients using the methods proposed, and how easy or difficult will this process be?

Can physicians deliver the proposed intervention messages in the time the investigators have proposed?

Can the phone counselor reach participants and accomplish the goals outlined for these calls?

Can the investigators obtain the data proposed and within the proposed time frame?

ELIGIBILITY:
Inclusion Criteria:

* child BMI ≥ 70th percentile for age and sex according to CDC Growth Tables
* child scheduled for an upcoming well child visit

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2006-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting and retaining families | Enrollment to 3-month followup

SECONDARY OUTCOMES:
Child weight (BMI) | Baseline and 3-months post
Parental perceptions of child weight | Baseline and 3-months post intervention
Satisfaction with intervention | 3-months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rona L Levy, MSW, PhD, MPH, Principal Investigator — University of Washington; Nancy Sherwood, PhD, Principal Investigator — Health Partners Research Foundation
Locations (2):
- United States (2):
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - University of Washington, Seattle, Washington